CLINICAL TRIAL: NCT06310304
Title: Relative Bioavailability of Ruxolitinib XR Tablets Compared With Ruxolitinib IR Tablets Administered Orally in Healthy Participants
Brief Title: A Study to Evaluate the Relative Bioavailability of Ruxolitinib Extended Release (XR) Tablets Compared With Ruxolitinib Immediate Release (IR) Tablets Administered Orally in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INCB18424-153
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Healthy Participants
Keywords: INCB018424; Ruxolitinib; Healthy Participants
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Dose Treatment A (Experimental): Ruxolitinib IR will be administered at protocol defined dose.
  Interventions: Drug: Ruxolitinib IR
- Cohort 1: Dose Treatment B (Experimental): Ruxolitinib XR will be administered at protocol defined dose.
  Interventions: Drug: Ruxolitinib XR
- Cohort 2: Dose Treatment A (Experimental): Ruxolitinib IR will be administered at protocol defined dose.
  Interventions: Drug: Ruxolitinib IR
- Cohort 2: Dose Treatment B (Experimental): Ruxolitinib XR will be administered at protocol defined dose.
  Interventions: Drug: Ruxolitinib XR

INTERVENTIONS:
Drug: Ruxolitinib IR — Tablet
  Other Names: INCB018424
  Arms: Cohort 1: Dose Treatment A; Cohort 2: Dose Treatment A
Drug: Ruxolitinib XR — Tablet
  Other Names: INCB018424
  Arms: Cohort 1: Dose Treatment B; Cohort 2: Dose Treatment B

SUMMARY:
This study is conducted to determine the Relative Bioavailability of Ruxolitinib XR Tablets Compared With Ruxolitinib IR Tablets Administered Orally in Healthy Participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Healthy adult participants aged 19 to 55 years at screening.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, at screening. Note: Only up to 25% of the participants in each cohort may be enrolled with a body mass index > 30 to ≤ 32.0 kg/m2.
* No clinically significant findings on screening evaluations (clinical, laboratory, and ECG).
* Ability to swallow and retain oral medication.
* Willingness to avoid pregnancy or fathering children based on the criteria below.

  * Male participants with reproductive potential must agree to take appropriate precautions to avoid fathering children (with at least 99% certainty) and not have a partner that is currently pregnant from screening through follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants who are WOCBP must have a negative serum pregnancy test at screening and a negative serum or urine pregnancy test at check-in before the first dose on Day -1 and must agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants of nonchildbearing potential (ie, surgically sterile with a hysterectomy and/or bilateral oophorectomy OR ≥ 12 months of amenorrhea and at least 51 years of age and FSH compatible with postmenopausal status) are eligible.

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening.
* History of cardiovascular, cerebrovascular, peripheral vascular or thrombotic disease or uncontrolled hypertension (blood pressure > 140/90 mmHg confirmed by repeat testing).
* Resting pulse < 45 bpm or > 100 bpm, confirmed by repeat testing.
* History or presence of an abnormal ECG before initial dose administration that, in the investigator's opinion, is clinically significant, such as a QTcF interval > 450 milliseconds.
* Presence of a malabsorption syndrome possibly affecting drug absorption (eg, Crohn's disease or chronic pancreatitis).
* Hemoglobin, WBC count, platelet count, or absolute neutrophil count less than laboratory lower limit of normal at screening or at check-in, confirmed by repeat testing.
* Hepatic transaminases (ALT and AST), ALP, or total bilirubin > 1.25 × the laboratory-defined ULN at screening and check-in, confirmed by repeat testing (except participants with Gilbert's disease, for which total bilirubin must be ≤ 2.0 × ULN).
* History of malignancy within 5 years of screening, with the exception of cured basal cell or squamous cell carcinoma of the skin, ductal carcinoma in situ, or Gleason 6 prostate cancer.
* Current or recent (within 3 months of screening) clinically significant gastrointestinal disease or surgery (including cholecystectomy) that could affect the absorption of study drug except that appendectomy will be allowed.
* Any major surgery within 4 weeks of screening.
* Donation of blood to a blood bank or in a clinical study (except a screening visit) within 4 weeks of screening (within 2 weeks for plasma only).
* Blood transfusion within 4 weeks of check-in.
* Chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment (includes latent treated tuberculosis).
* Positive test for hepatitis B virus, HCV, or HIV. Participants whose results are compatible with prior immunization or immunity due to infection for hepatitis B may be included at the discretion of the investigator.
* History of alcoholism within 3 months of screening.
* Positive urine or breath test for ethanol or positive urine screen for drugs of abuse that are not otherwise explained by permitted concomitant medications or diet.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with another investigational medication or current enrollment in another investigational drug Protocol.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with an inducer or inhibitor of cytochrome P450 3A4, P-glycoprotein, or breast cancer resistance protein.
* Current use of prohibited medication.
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) deemed clinically relevant by the investigator.
* Known hypersensitivity or severe reaction to ruxolitinib or any excipients of ruxolitinib.
* Inability to undergo venipuncture or tolerate venous access.
* Inability or unlikeliness of the participant to comply with the dose schedule and study evaluations, in the opinion of the investigator.
* Use of tobacco- or nicotine-containing products within 1 month of screening and throughout the study.
* Use of prescription drugs within 14 days of study drug administration or nonprescription medications/products (including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations) within 7 days of study drug administration and throughout the study except for permitted medications during the study.
* Women who are pregnant or breastfeeding.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* eGFR < 90 mL/min/1.73 m2 based on the site's standard formula.
* Any condition that would jeopardize the safety of the participant or compliance with the Protocol.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
INCB018424 pharmacokinetic (PK) in Plasma | Up to Day 22
  INCB018424 concentration in plasma.

SECONDARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | Up to Day 55
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Additional INCB018424 pharmacokinetic (PK) in Plasma | Up to Day 22
  Additional INCB018424 concentration in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Celerion, Inc, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No